CLINICAL TRIAL: NCT02778490
Title: Effects of Sleeve Gastrectomy on Calcium Metabolism and the Skeleton
Status: Completed | Type: Observational
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: University of California, San Francisco (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Anne Schafer, Assistant Professor of Medicine and of Epidemiology and Biostatistics; Staff Physician, San Francisco Veterans Affairs Medical Center
Other Study IDs: R01DK107629 (NIH); R01DK107629 (NIH)
Record Dates: First submitted 2016-05-15; First posted 2016-05-20 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Calcium Metabolism Disorders; Morbid Obesity
Keywords: sleeve gastrectomy, bariatric surgery
MeSH Terms: conditions — Calcium Metabolism Disorders; Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, urine
Oversight: Data Monitoring Committee: No

SUMMARY:
In this pre-post observational study, the investigators will enroll and follow a cohort of about 50 adults undergoing sleeve gastrectomy surgery for weight loss. Pre-operatively and at 6 and 12 months post-operatively, the investigators will use state-of-the-art metabolic and imaging techniques to evaluate calcium metabolism and skeletal health. Specific outcomes include intestinal calcium absorption capacity, bone mineral density (BMD) assessed by dual-energy X-ray absorptiometry (DXA) and quantitative computed tomography (QCT), and bone structure assessed by QCT and high-resolution peripheral QCT (HR-pQCT).

DETAILED DESCRIPTION:
Obesity is a chronic disease of staggering proportions. Because weight loss through diet and exercise is difficult to attain and maintain, there is escalating interest in surgical weight loss procedures, including Roux-en-Y gastric bypass. Gastric bypass results in marked and durable weight loss and improvement in comorbidities in the general population and in our veteran patients. However, growing evidence indicates that gastric bypass can have negative effects on the skeleton, increasing bone turnover and decreasing bone mineral density (BMD). This is of critical concern given the tremendous impact of osteoporosis and fracture in both men and women. Vitamin D deficiency due to obesity and post-surgical malabsorption may partially explain the decline in bone mass observed after gastric bypass. Other factors are likely involved as well, such as non-vitamin D-mediated calcium malabsorption, signals related to decreased skeletal loading, and changes in fat-secreted hormones or estrogen (due to changes in fat mass and body composition).

We will characterize the effects of gastric bypass on calcium metabolism and the skeleton in a cohort of 80 men and women whose serum 25-hydroxyvitamin D levels are supplemented and maintained at ≥30 ng/mL. First, we will test the hypothesis that intestinal calcium absorption is impaired following gastric bypass, even in the setting of vitamin D sufficiency. We will do this by measuring fractional calcium absorption pre-operatively and 6 months post-operatively using dual stable isotopic tracers (Aim 1). Then, we will test the hypothesis that gastric bypass results in decreased BMD and in structural changes associated with impaired skeletal strength. We will do this by performing dual-energy X-ray absorptiometry (DXA), quantitative computed tomography (QCT), and high-resolution peripheral QCT (HR-pQCT) pre-operatively and 6 and 12 months post-operatively (Aim 2). QCT and HR-pQCT are advanced imaging techniques that have distinct advantages over standard methods but have not yet been applied to this population. Finally, we will assess body composition changes by anthropometry, DXA, and QCT, and changes in fat-secreted hormones, and we will evaluate the relationship between changes in skeletal parameters and changes in body composition and hormones (Aim 3). This research is expected to impact the clinical care of gastric bypass patients by helping to shape recommendations about post-operative nutrition, BMD screening, and potential therapy.

As an ancillary study aim (Aim 4), we will assess vertebral bone marrow fat pre- and post-operatively in a subgroup of participants, and we will evaluate the relationships between change in vertebral bone marrow fat, changes in body composition and fat-secreted hormones, and changes in skeletal parameters. The participants in this subgroup will have the option of undergoing additional knee tissue composition evaluation, allowing us to evaluate the relationship between weight loss and change in knee health. In order to develop and refine the magnetic resonance (MR) sequences we will use for Aim 4, we will scan a small group of healthy controls at baseline and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Women and men 25 to 70 years old scheduled to undergo sleeve gastrectomy

Please note that the investigators are unable to provide sleeve gastrectomy; rather, potential participants must already be planning the procedure with their surgeons.

Exclusion Criteria:

* Perimenopausal women, defined as last menses >3 months but < 5 years ago
* Known intestinal malabsorption (e.g., celiac disease, short gut syndrome, prior intestinal surgery)
* Prior bariatric surgery
* Use of medications known to impact bone and mineral metabolism, including use of a bisphosphonate or teriparatide in the last year or for >12 months ever; current calcitonin; prednisone >5 mg daily or the equivalent glucocorticoid for >10 days in the last 3 months; a current thiazolidinedione (TZD); an aromatase inhibitor; androgen deprivation therapy; an antiepileptic agent known to alter hepatic vitamin D clearance; or thyroid hormone replacement with current thyroid stimulating hormone < 0.1 milli-international units per liter
* Disease known to affect bone (e.g., primary hyperparathyroidism, Pagets disease, clinically significant liver disease)
* Illicit drug use or alcohol use >3 drinks/day
* Serum calcium >10.2 mg/dL or calculated creatinine clearance < 30 mL/min
* Weight >350 pounds (the maximum weight limit of the QCT scanner) at the time of the pre-operative QCT scan

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese men and women undergoing sleeve gastrectomy surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2021-11-28 (Actual); Study Completion 2021-11-28 (Actual)

PRIMARY OUTCOMES:
Change in intestinal fractional calcium absorption | 6 months
  The investigators will determine whether there is a change in intestinal calcium absorption, assessed using the dual stable isotopes Ca-43 and Ca-44 in the setting of robust vitamin D status, following sleeve gastrectomy.

SECONDARY OUTCOMES:
Percentage change in spinal volumetric bone mineral density | 12 months
  The investigators will define the effects of sleeve gastrectomy on spinal volumetric bone mineral density, assessed by quantitative computed tomography (QCT).
Percentage change in volumetric bone mineral density at the distal tibia | 12 months
  The investigators will define the effects of sleeve gastrectomy on total volumetric bone mineral density at the distal tibia, assessed by high-resolution peripheral quantitative computed tomography (HR-pQCT).
Percentage change in cortical porosity at the distal tibia | 12 months
  The investigators will define the effects of sleeve gastrectomy on cortical porosity at the distal tibia, assessed by high-resolution peripheral quantitative computed tomography (HR-pQCT).

OTHER OUTCOMES:
Percentage change in spinal volumetric bone mineral density by QCT | 6 months
Percentage change in volumetric bone mineral density at the distal tibia by HR-pQCT | 6 months
Percentage change in cortical porosity at the distal tibia by HR-pQCT | 6 months
Percentage changes in cortical and trabecular volumetric bone mineral density and microstructural parameters at the radius and tibia by HR-pQCT | 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Schafer, MD, Principal Investigator — San Francisco VA Medical Center
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No